CLINICAL TRIAL: NCT03774355
Title: A Randomized, Open-label, Single, 2x2 Crossover Study to Compare the Safety and Pharmacokinetics of "CG1801" and "CGL1802" in Healthy Volunteers
Brief Title: Study to Compare Safety and Pharmacokinetics of "CG1801" and "CGL1802" in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CG100649-1-07
Record Dates: First submitted 2018-12-09; First posted 2018-12-12 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CG1801 (Experimental): Dosing 'CG1801' followed by dosing 'CGL1802'
  Interventions: Drug: CG1801
- CGL 1802 (Experimental): Dosing 'CGL1802' followed by dosing 'CG1801'
  Interventions: Drug: CGL1802

INTERVENTIONS:
Drug: CG1801 — Administration CG1801 2mg single dose in phase 1 and Administration CGL1802 2mg single dose phase 2.
  Arms: CG1801
Drug: CGL1802 — Administration CGL1802 2mg single dose in phase 1 and Administration CG1801 2mg single dose phase 2
  Arms: CGL 1802

SUMMARY:
The objective of this open-label, randomized, 2*2 crossover study is to compare the safety and Pharmacokinetics CG1801 and CGL1802 in Healthy Volunteers.

DETAILED DESCRIPTION:
Healthy volunteers are administrated single-dose over the period I and II (crossover) of CGL1802(Polmacoxib 2mg Tablet) and CG1801(Polmacoxib 2mg capsule) Every time before and after each medication, pharmacokinetic (PK) parameters and safety of CGL1802 and CG1801 is performed using a blood sample and conducting some tests (vital signs, physical exam, ECG, laboratory test, etc.) respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥ 19 years and ≤ 50 years
2. Without inborn or chronic disease and no symptoms in physical examination
3. BMI(Body Mass Index) result ≥ 18kg/m 2 and ≤ 30kg/m2
4. Adequate clinical laboratory test results as evidenced by Hematology, Hemostasis, Biochemistry, Urinalysis, Serology and so on
5. After taking a rest in sitting position for 5 minutes, subjects who have blood pressure (90 mmHg ≤ Systolic BP ≤ 139 mmHg, and 60 mmHg ≤ Diastolic BP ≤ 89 mmHg)
6. Subject who understand the objective, method of the study and the characteristics of investigational drug and expected adverse events and provide written informed consent prior to study participation
7. Negative pregnancy test(hCG) and agree to contraception during the trial

Exclusion Criteria:

1. History of hypersensitivity to investigational products
2. History of hypersensitivity or allergic reaction to sulfonamide.
3. Patients with a history of asthma, acute rhinitis, nonspecific polyps, angioedema, urticaria or allergic reactions to aspirin or other nonsteroidal anti- inflammatory analgesics (including COX-2 inhibitors)
4. Uncontrolled hypertension (over the Systolic BP 140 mm Hg or Diastolic BP 90 mmHG)
5. Edema or Fluid retention
6. AST / ALT > 1.5 times the normal range including additional and Screening blood tests before randomization.
7. MDRD < 60mL / min / 1.73m2 including additional and Screening blood tests before randomization.
8. Patient with an active peptic ulcer or gastrointestinal bleeding
9. Patient with inflammatory intestinal disease such as Crohn's disease or ulcerative colitis
10. Patient with Congestive Heart Failure (NYHA II - IV)
11. Established ischemic heart disease patients, peripheral arterial diseases, and/or brain vascular diseases patient
12. Patient performed CABG within 30 days prior to the first administration of the investigational drug
13. Patient has hyperkalemia
14. Patient has blood coagulation disorder or administration the anticoagulant
15. Patient with gastrointestinal related disease or gastrotomy history (except appendicitis or hernia surgery) that may affect the absorption of the investigational drug.
16. Patient participated in any other clinical trials or Bio-equivalence studies within 90 days prior to the screening visit.
17. Patient donated whole blood within 60 days, donated blood component within 14 days, or received blood transfusion within 30 days prior to the first administration of the investigational drug.
18. Taken medications like barbital or herbal medicines within 30 days or taken Over The Counter medicines within 7 days prior to the first administration of the investigational drug that may affect the clinical trial
19. Over smokers (tobacco > 20 cigarettes/ days) within 30 days prior to Screening visit or patient cannot quit smoking during and until the end of the clinical trial after signed the Informed Consent Form to participate the clinical trial.
20. Excessive Alcohol consumer 30 days prior to Screening visit or cannot quit drinking alcohol during and until the end of the clinical trial after signed the Informed Consent Form to participate the clinical trial.
21. Excessive caffeine consumer (> 5 drinks/ day)
22. Breast Feeding woman
23. Patient cannot accept medically acceptable contraception during and until the clinical trial.
24. Any other reasons or situations that the investigator decides the patient is not eligible to participate the clinical trial.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Area Under Curve [AUC]last of polmacoxib AUClast of polmacoxib AUClast of polmacoxib AUClast of polmacoxib | Day1 pre-dose and each of the post-doses of each of the 2 treatment periods in CG1801 and CGL1802 Group.
  Area Under Curve [AUC]last of CGL1802 will be evaluated
Maximum Plasma Concentration [Cmax] of polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
  Maximum Plasma Concentration [Cmax] of CGL1802 will be evaluated

SECONDARY OUTCOMES:
Area Under Curve [AUC]last of polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
Maximum Plasma Concentration [Cmax] of polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
AUCinf of polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
Time to maximum plasma concentration [Tmax] of polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
t1/2 of polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
clearance [CL/F] of Polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.
Volume of distribution [Vd/F] of Polmacoxib | Day1 pre-dose and each of the post-doses of the 2 treatment periods in CG1801 and CGL1802 Group.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea